CLINICAL TRIAL: NCT01672918
Title: Use of Fluorodeoxyglucose Positron Emission Tomography With Computed Tomography for the Evaluation of Autoimmune Lymphoproliferative Syndrome Lymphadenopathy Suggestive of Lymphoma
Brief Title: Fluorodeoxyglucose Imaging Studies to Detect Lymphoma
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120184; 12-I-0184
Record Dates: First submitted 2012-08-23; First posted 2012-08-27 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2015-02-27

CONDITIONS: Autoimmune Lymphoproliferative Syndrome; Lymphoma
Keywords: PET/CT; Lymphoma; Lymphadenopathy; ALPS
MeSH Terms: conditions — Autoimmune Lymphoproliferative Syndrome; Lymphoma; Lymphadenopathy

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Autoimmune lymphoproliferative syndrome (ALPS) is a genetic disorder of the lymph system. People with ALPS often have swollen lymph nodes, especially in the neck and armpit. They also have a much higher risk of developing lymphoma. It is not always easy to determine whether the swollen lymph nodes are caused by ALPS or by lymphoma. Researchers want to see whether different imaging studies can show the difference between ALPS and lymphoma. The studies used will be positron emission tomography (PET) and computed tomography (CT). Researchers will use a drug called fluorodeoxyglucose (FDG) to look at the lymph nodes.

Objectives:

- To see how well imaging studies can distinguish between swollen lymph nodes caused by ALPS or by lymphoma.

Eligibility:

* Individuals must be 5 years of age or older and enrolled on the National Institutes of Health natural history study of ALPS.
* Participants should either have lymphoma or have symptoms that suggest possible lymphoma.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Participants will have an FDG-PET/CT scan. It will be performed according to standard procedures.
* If the results of the scan do not show lymphoma, participants will stay on the study for 1 year for clinical follow up. They may have a second FDG-PET/CT scan if there is a change in symptoms. Such changes include further enlargement of lymph nodes, unexplained fevers, or weight loss.
* If the results of the scan show evidence of new or worsening lymphoma, treatment on this study will end. Further tests based on clinical symptoms, including a lymph node biopsy, may be done under the ALPS natural history study to rule out or make a diagnosis of lymphoma.

DETAILED DESCRIPTION:
The Autoimmune Lymphoproliferative Syndrome (ALPS) is an inherited disorder associated with defective lymphocyte apoptosis, which is clinically characterized by prominent nonmalignant lymphadenopathy, hepatosplenomegaly, and overt autoimmune diseases such as hemolytic anemia, autoimmune thrombocytopenia, and neutropenia. Additionally, ALPS patients have a significantly increased risk of developing non-Hodgkin lymphoma (NHL) and Hodgkin lymphoma (HL). The diagnosis of lymphoma is particularly troublesome in ALPS because many ALPS manifestations overlap with clinical features suggestive of lymphoma. Therefore, individuals with ALPS may undergo repeated biopsies during the course of the disease. Fluorodeoxyglucose positron emission tomography combined with computed tomography (FDG-PET/CT) is a noninvasive test that may help us discriminate benign from malignant lymphadenopathy in patients with ALPS.

For patients with ALPS and clinical symptoms suggestive of lymphoma, such as a sudden increase in focal lymphadenopathy and/or systemic B symptoms associated with lymphoma, we want to investigate whether FDG-PET/CT is useful in determining a plan of action by assisting in locating the most active lymph node and determining whether a surgical biopsy is warranted. Under this protocol, FDG-PET/CT scans will be done to rule out lymphoma. A lymph node biopsy may be necessary to determine the pathology of the lymph node and will not be done for research purposes alone.

ELIGIBILITY:
* INCLUSION CRITERIA:

To qualify for enrollment, patients must meet all of the following:

1. Fulfill current criteria for the diagnosis of ALPS, which includes documented chronic nonmalignant lymphadenopathy and/or splenomegaly, and either greater than or equal to 1.5% T-cell receptor alpha/beta+ DNTs in the peripheral blood or confirmed RAS mutation with or without elevated alpha/beta DNTs.
2. Be enrolled in ALPS natural history protocol #93-I-0063.
3. Have 1 or more of the following:

   1. Sudden enlargement of at least 1 lymph node or group of lymph nodes over baseline.
   2. Systemic symptoms suspicious for lymphoma (i.e., loss of weight, loss of appetite, fatigue, night sweats, fever, and pruritus).
   3. A histologically proven diagnosis of lymphoma or other malignancy.
4. Be 5 years of age or older.

EXCLUSION CRITERIA:

Patients will be excluded if any of the following is present:

1. Concurrent proven infection or inflammatory disease (e.g., sarcoidosis), which itself often shows increased FDG uptake by PET and which could interfere with the interpretation of study results.
2. Hyperglycemia (regardless of etiology) determined by fasting glucose of >200 mg/dL
3. Weight in excess of 400 lb, which will exceed the weight limit for the scanner table.
4. Pregnancy or breast-feeding. For women of childbearing potential, a negative urine or serum pregnancy test is required within 24 hours prior to an FDG-PET/CT scan.

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08-06; Study Completion 2015-02-27

CONTACTS AND LOCATIONS:
Overall Officials: V. Koneti Rao, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)

REFERENCES:
- [Background] Sneller MC, Wang J, Dale JK, Strober W, Middelton LA, Choi Y, Fleisher TA, Lim MS, Jaffe ES, Puck JM, Lenardo MJ, Straus SE. Clincal, immunologic, and genetic features of an autoimmune lymphoproliferative syndrome associated with abnormal lymphocyte apoptosis. Blood. 1997 Feb 15;89(4):1341-8. PMID 9028957
- [Background] Straus SE, Sneller M, Lenardo MJ, Puck JM, Strober W. An inherited disorder of lymphocyte apoptosis: the autoimmune lymphoproliferative syndrome. Ann Intern Med. 1999 Apr 6;130(7):591-601. doi: 10.7326/0003-4819-130-7-199904060-00020. PMID 10189330
- [Background] Avila NA, Dwyer AJ, Dale JK, Lopatin UA, Sneller MC, Jaffe ES, Puck JM, Straus SE. Autoimmune lymphoproliferative syndrome: a syndrome associated with inherited genetic defects that impair lymphocytic apoptosis--CT and US features. Radiology. 1999 Jul;212(1):257-63. doi: 10.1148/radiology.212.1.r99jl40257. PMID 10405750